CLINICAL TRIAL: NCT06090149
Title: Telemedical Assistance in Automatic Titration of Oxygen for Intensive Care Patients
Acronym: Smartassistant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E1.1.1.1/21/A/082
Record Dates: First submitted 2023-09-11; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Obesity Hypoventilation Syndrome (OHS); Chronic Obstructive Lung Disease; Interstitial Lung Disease; Pneumonia
Keywords: Telemedicine; Smart assistant
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Pneumonia

STUDY DESIGN:
Intervention Model Description: Pre/post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP/APAP INTERVENTION WITH AND WITHOUT OXYGEN SUPPORT (Experimental): Patients in this group will be selected from the Sleep Disorder Center database for printing data on hypoxemia below 90% during the night and for treatment received (CPAP/APAP and/or oxygen therapy). And from available data in PSCUH data systems on patient diagnoses, previous results of studies (results of blood gas tests), and recommended treatments on hospital and outpatient disease cards, which will include indications of possible chronic hypoxemia. The selected patients will be called (telephone visit) and, if agreed, will be scheduled for study time. Consequently, if the consent questionnaire was signed, a study will be launched following an evaluation of the inclusion and exclusion criteria.
  Interventions: Device: PHASE 1 Lowenstein medical BiLevel Prisma 25ST device: withount oxygen support.; Device: PHASE 2. Continous/Bilevel positive airway presure with additional oxygen support by Devilbiss 525 KS oxygen concentrator

INTERVENTIONS:
Device: PHASE 1 Lowenstein medical BiLevel Prisma 25ST device: withount oxygen support. — The patient will be invited to enter the study's first phase using the Lowenstein medical BiLevel Prisma 25ST device without additional oxygen support. The study will be conducted within 1-3 days. If patients fail to achieve proper blood oxygen saturation without oxygen supplementation, patient will be selected to proceed to the next step - oxygen-enriched positive airway pressure intervention
  During monitoring TA, RR, HR, SpO2, as well as CO2 in both exhales/inhales and transcutaneous positions will be measured by Lowenstein Medical Sonata and Sentec device.
Device: PHASE 2. Continous/Bilevel positive airway presure with additional oxygen support by Devilbiss 525 KS oxygen concentrator — The patient will be invited to enter the third phase of the study with rapid oxygen titration. Titration occurs in an inpatient department where the patient is connected to the Lowenstein medical BiLevel Prisma 25ST device with oxygen support during the daytime. As part of the study, the patient will be supplied with oxygen by Devilbiss 525 KS oxygen concentrator at a dosing interval of 1-10 L/min. Every 2 hours oxygen support will be increased by 2L/min.
  During monitoring TA, RR, HR, SpO2, and CO2 in both exhales/inhales and transcutaneous positions will be measured by Lowenstein Medical Sonata and Sentec device.

SUMMARY:
The goal of this clinical trial is to clinically validate a system for the monitoring of patients' respiratory function and automated oxygen treatment proposal using non-invasive ventilation devices in the treatment of intensive care patients with acute or chronic lung diseases exacerbations. Participants clinical parameters will be monitored and samples will be sent to a clinical laboratory for analysis (arterial blood pressure, heart rate, and respiratory rate will be continuously recorded, and FeO2 and CO2 will be measured with the help of an additional sensor).

DETAILED DESCRIPTION:
This prospective experimental study is conducted in Pauls Stradins Clinical University Hospital (PSCUH) and Sleep Disease Center in Riga, Latvia. The study includes patients with respiratory failure and hypoxemia to whom NIV is indicated.

Participants clinical parameters are monitored and samples will be sent to a clinical laboratory for analysis.

Initial ventilation parameters will be defined by the clinician who performs the experiment.

During the validation phase, the investigators will obtain clinicians' final decision on the changes of the ventilation system parameters and compare it to our module proposal. That way it would be possible to estimate if the system is ready for the next step - fully automated closed-loop ventilation system development.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent to participate in the study;
* aged over 18 years;
* patients hospitalized with acute respiratory failure (indication to NIV therapy) with restrictive or obstructive lung disease

Exclusion Criteria:

* refusal to participate further in the study;
* age under 18 years;
* pregnancy;
* the patient is contraindicated for non-invasive lung ventilation
* during the study, the patients condition worsens in such a way that an active one is required medical intervention or continuation of the study may worsen the patients condition;
* complications related to NIV therapy or claustrophobia;
* chronic obstructive pulmonary disease and obstructive sleep apnea without documented hypoxemia (Sp02 and Sa02 > 94%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 11 months
  The change in the Apnea-Hypopnea Index (AHI) within oxygen titration will be measured pre-interventionally and during the intervention.
Transcutaneous CO2 partial pressure (tcCO2) | 11 months
  The change in transcutaneous CO2 partial pressure (mmHg) within oxygen titration and the time spent within an acceptable CO2-interval measured pre-interventionally and during the intervention.
Blood Oxygen Saturation (SpO2) | 11 months
  Evaluation will include the difference in blood Oxygen Saturation (SpO2%) pre-interventionally and during the intervention.
Blood pressure (TA) | 11 months
  Evaluation will include the difference in the blood pressure (mmHg) measures pre-interventionally and during the intervention.
Respiratory rate (RR) | 11 months
  Evaluation will include the difference in the respiratory rate (xmin) measures pre-interventionally and during the intervention.
Heart rate (HR), | 11 months
  Evaluation will include the difference in the heart rate (xmin) pre-interventionally and during the intervention.
Upper airway Carbon dioxide levels (CO2) | 11 months
  The change in CO2 (mmHg) within oxygen titration will be measured pre-interventionally and during the intervention.

SECONDARY OUTCOMES:
adverse events description | 11 months
  all adverse events recorded by investigators in the CRF

CONTACTS AND LOCATIONS:
Locations (1):
- Pauls Stradins Clinical Univeristy Hospital, Riga, Latvia